CLINICAL TRIAL: NCT02648633
Title: A Pilot Study to Evaluate the Feasibility of the Combined Use of Stereotactic Radiosurgery With Nivolumab and Concurrent Valproate in Patients With Recurrent Glioblastoma
Brief Title: Stereotactic Radiosurgery With Nivolumab and Valproate in Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmaceutical company (BMS) would no longer provide nivolumab for the study, so the study was terminated early.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Benjamin Purow, MD, Professor of Neurology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18574; CA209-378 (Other: University of Virginia)
Record Dates: First submitted 2015-12-16; First posted 2016-01-07 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma
Keywords: Brain Cancer; Immunotherapy; Nivolumab; Radiosurgery; Gamma Knife
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Radiosurgery; Nivolumab; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab & Valproate Following G.K. (Experimental): Subjects will begin a valproate regimen prior to undergoing stereotactic radiosurgery (gamma knife) on a single lesion. Following the surgery, subjects will receive nivolumab every 2 weeks and daily valproate.
  Interventions: Radiation: Stereotactic Radiosurgery; Drug: Nivolumab; Drug: Valproate

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Subjects will receive a single large dose of radiation to one or more lesions.
  Other Names: Gamma Knife Radiosurgery
Drug: Nivolumab — 3 mg/kg of nivolumab will be administered through IV infusion every two weeks following stereotactic radiosurgery.
  Other Names: Opdivo
Drug: Valproate — Subjects will begin regimen of valproate prior to radiosurgery and continue to receive therapy concurrently with nivolumab. Subjects will receive valproate daily with a target serum level of 75-100 μg/ml.
  Other Names: Valproic Acid; Sodium Valproate; Divalproex Sodium

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the immunotherapeutic agent nivolumab given in combination with gamma knife therapy and valproate in patients with recurrent glioblastoma, a common and lethal type of brain cancer.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors have the potential to treat a wide range of diverse cancers. Of particular interest to researchers is the PD-1 receptor-ligand interaction, a major pathway that many cancers hijack in order to suppress immune control. Anti-PD-1 antibodies such as nivolumab show a strong potential to treat many types of cancers including glioblastoma, the most common and most lethal brain cancer.

This study will examine a means of further focusing immune response on glioblastoma by combining stereotactic "gamma knife" radiosurgery with nivolumab. The rationale behind this intervention is that the radiation therapy will enhance immune response rate by providing additional tumor antigens from dying cells. Additionally, a study from investigators at Johns Hopkins indicates that histone deacetylase (HDAC) inhibitors may boost the anti-cancer efficacy of PD-1 antibodies like nivolumab. Valproate, a class I HDAC inhibitor, will be used concurrently with nivolumab with the goal of enhancing the effects of both the nivolumab and the radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignant, recurrent glioblastoma or gliosarcoma
* Subject must have adequate organ function
* Subject must still be able to care for most of his or her personal needs

Exclusion Criteria:

* Subject is pregnant
* Subject has extracranial metastatic or leptomeningeal disease
* Subject has an additional malignancy that is progressing or requires active treatment, exceptions being basal cell and squamous cell carcinomas of the skin, indolent prostate cancer, chronic lymphocytic leukemia, or in situ cervical cancer
* Subject has received chemotherapy, biological therapy, or had surgery 4 weeks prior to beginning the study
* Subject has had radiation therapy within 10 weeks prior to entering beginning the study
* Subject has had prior therapy with bevacizumab
* Subject has had previous treatment with carmustine wafer except when administered as first-line treatment no less than six months prior to beginning the study
* Subject requires escalating supraphysiologic doses of corticosteroids greater than 2 mg of dexamethasone or an equivalent
* Active autoimmune disease requiring systemic treatment within the past 3 months or any syndrome that requires immunosuppressive agents
* Interstitial lung disease or active, non-infectious pneumonitis
* Evidence of greater than Grade 1 CNS hemorrhage or greater than Grade 3 venous thromboembolism
* History of uncontrolled cardiac disease
* Subject unable or unwilling to have a head contrast enhanced MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Feasibility based on number of subjects who complete 4 doses of nivolumab | At 3 months following radiosurgery
  Feasibility of the radiosurgery and drug combination will be determined based on the number of subjects who complete at least 4 doses of nivolumab.
Incidence of adverse events | From the beginning of treatment until no sooner than 30 days following the last study treatment
  Safety will be assessed by imaging of necrosis, incidence and severity of adverse events, changes in laboratory findings, physical examinations, vital signs, and the number of discontinuations due to adverse events.

SECONDARY OUTCOMES:
Clinical Response Rate | From the beginning of treatment until documented disease progression or date of death, assessed up to 48 months.
  Response to therapy will be evaluated by means of RANO criteria.

OTHER OUTCOMES:
Incidence of Pseudoprogressions | From the beginning of treatment until documented disease progression or date of death, assessed up to 48 months.
  Pseudoprogression, the transient increase in apparent tumor size, will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Purow, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No